CLINICAL TRIAL: NCT00906594
Title: Additive Intra-ocular Pressure Reduction Effect of Fixed Combination of Maleate Timolol 0.5%/Dorzolamide 2% on Monotherapy With Latanoprost in Patients With Elevated Intra-ocular Pressure: a Prospective, Four-week, Open-label, Randomized, Controlled Clinical Trial.
Brief Title: Additive Intra-ocular Pressure Reduction Effect of Fixed Combination of Maleate Timolol 0.5%/Dorzolamide 2% on Monotherapy With Latanoprost in Patients With Elevated Intra-ocular Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Marcelo Hatanaka, Head, Glaucoma Service, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Merck-USP-01; NCT00766922 (obsolete NCT alias)
Record Dates: First submitted 2009-05-18; First posted 2009-05-21 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Latanoprost

ARMS (2):
- Latanoprost (Active Comparator): Latanoprost mono therapy
  Interventions: Drug: latanoprost
- Latanoprost + Fixed combination (Experimental): Latnoprost + Fixed combination
  Interventions: Drug: latanoprost

INTERVENTIONS:
Drug: latanoprost

SUMMARY:
The purpose of this study is to evaluate the additive effect of dorzolamide/timolol fixed combination in patients undergoing monotherapy with latanoprost.

ELIGIBILITY:
Inclusion Criteria:

All patients were at least 18 years old, with unilateral or bilateral open-angle glaucoma (defined as IOP > 21 mmHg, mean of three consecutive measurements, at any time during the day, at the moment of glaucoma diagnosis) or ocular hypertension (IOP> 25 mmHg, mean of three consecutive measurements, at anytime during the day, at the moment of diagnosis). Glaucoma was defined as a reproducible glaucomatous visual field defect based on GHT outside normal limits and/or PSD lower than 0,5% or glaucomatous changes of the optic disc associated to elevated IOP. A visual acuity (ETDRS) of 20/80 or better was required for randomization.

Exclusion Criteria:

Included woman of childbearing potential, pregnancy, systemic contra-indication to beta-blocker therapy, argon laser trabeculoplasty three months before screening visit, any history of filtering surgery, ocular surgery or uveitis three months before screening visit, hypersensitivity to any compound of the study drugs, concomitant use of any experimental drug, any condition in which treatment with beta-blocker is contraindicated or any other abnormal and/or ocular condition or symptom that would prevent study participation, according to the judgment of the investigator. The use of systemic beta-blocker, if needed, was allowed and not considered an exclusion criterion. Latanoprost non-responders defined as lower than 15% IOP reduction after run-in period with latanoprost monotherapy were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
additional IOP reduction obtained with cosopt in addition to xalatan | 4 week

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil